CLINICAL TRIAL: NCT04161027
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Study to Assess Efficacy and Safety of Pregabalin in Willis-Ekbom Disease/Restless Legs Syndrome
Brief Title: RCT for Pregabalin in Restless Legs Syndrome in South Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ki-Young Jung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1903-121-1021
Record Dates: First submitted 2019-11-06; First posted 2019-11-13 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Restless Legs Syndrome
Keywords: Restless legs syndrome; pregabalin; Willis-Ekbom disease
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pregabalin

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, multicenter clinical trial. Study subjects will be recruited from 4 medical centers in South Korea.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin 75mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Pregabalin 75mg — Pregabalin 75 mg capsule
  Arms: Pregabalin
Drug: Placebos — Placebo capsule
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, multicenter clinical trial is designed to to assess the treatment efficacy and tolerability of pregabalin in patients with idiopathic restless legs syndrome in South Korea.

DETAILED DESCRIPTION:
Objectives: To assess the treatment efficacy and tolerability of pregabalin in patients with idiopathic restless legs syndrome (RLS) in South Korea.

Study Design: A randomized, double-blind, placebo-controlled, multicenter clinical trial Study period: total 14 weeks: 2 weeks for placebo run in period and 12 weeks treatment after randomization (titration for 4 weeks and maintenance for 8 weeks).

Subjects: a total number of 100 participants (randomly assigned 1:1 to pregabalin or placebo). The sample number was calculated based on a superiority design, 1-sided, alpha 0.05 with power 80% and drop rate 10%.

Inclusion criteria: adults aged between 19-80 and diagnosed with idiopathic RLS with IRLS score of 15 or more.

Exclusion criteria: Secondary RLS; serum ferritin < 10 μg/L or history of oral iron therapy within 3 months or intravenous iron therapy within 1 year; severe comorbid medical or psychiatric disorders; history of pregabalin or gabapentin treatment within 3 months; other comorbid sleep disorders or shift workers.

Treatment schedule and dose

- Placebo responders, who showed a decrease of IRLS score of 40% or more, are excluded before randomization. Subjects will randomly assigned to receive either pregabalin or placebo with a 1:1 allocation. A starting dose is 75 mg/day for 2 weeks (taken 1-2 hours before habitual bedtime). At the visit of 2 weeks and 4 weeks, a dose can be titrated by 75-150 mg according to the response and tolerability. A dose ranging 75-300 mg per day will be maintained for 8 weeks.

Primary outcome: changes in IRLS score after 12-week treatment. Secondary outcomes: remission rate (decrease in IRLS score of 50% or more), CGI (clinical global impression)-improvement, changes in 10-cm visual analog scale (VAS), RLS-6, PSQI (pittsburgh sleep quality index), ISI (insomnia severity index), Johns Hopkins RLS QoL after 12-week treatment.

Statistical analysis: ANCOVA for changes in IRLS score with a baseline IRLS score as a covariate.

Tolerability: Safety profiles and Liverpool Adverse Event Profile (LAEP) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* IRLS (international restless legs scale) score ≥ 15
* RLS symptom occurring ≥ 3 times/week and persisting over ≥ 6 months
* Drug-naive patients or those who stop taking RLS drugs for ≥ 1 week before screening

Exclusion Criteria:

* Secondary RLS (including iron deficiency anemia, pregnancy, chronic kidney disease [eGFR < 60 mL/min/1.73 m2], peripheral neuropathy, others)
* Serum Ferritin < 10 μg/L or history of oral iron therapy within 3 months or intravenous iron therapy within 1 year
* Severe comorbid medical or psychiatric disorders
* history of pregabalin or gabapentin treatment within 3 months
* High risk of obstructive sleep apnea by STOP-BANG questionnaire
* Other comorbid sleep disorders or shift workers
* Hypersensitivity to pregabalin
* Galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
International restless legs scale score | Baseline (week 0) and post-treatment (week 12)
  Changes in International restless legs scale (IRLS) score after 12-week treatment. IRLS is used to assess the severity of patient's RLS symptoms. A total score ranges from 0 to 40 and higher scores mean more severe symptoms. Therefore, greater differences in IRLS scores between baseline and post-treatment mean a better outcome.

SECONDARY OUTCOMES:
Remission rate | Baseline (week 0) and post-treatment (week 12)
  A proportion of patients who showed a decrease in IRLS score of 50% or more after treatment. Higher scores mean a better outcome.
CGI (clinical global impression)-improvement | Post-treatment (week 12)
  The amount of RLS symptom improvement measured by physicians. CGI-improvement is a 7-point scale and rated as 1 (Very much improved), 2 (Much improved), 3 (Minimally improved), 4 (No change), 5 (Minimally worse), 6 (Much worse), and 7 (Very much worse).
10-cm visual analog scale (VAS) | Baseline (week 0) and post-treatment (week 12)
  Changes in 10-cm VAS after 12-week treatment. A VAS score ranges from 0 (no symptoms) to 10 (very severe symptoms).
Restless legs syndrome (RLS)-6 | Baseline (week 0) and post-treatment (week 12)
  Changes in RLS-6 scores after 12-week treatment. A RLS-6 consists of 6 questions for RLS symptoms and a total score ranges from 0 (no symptoms) to 60 (very severe symptoms).
PSQI (pittsburgh sleep quality index) | Baseline (week 0) and post-treatment (week 12)
  Changes in PSQI scores after 12-week treatment. A total PSQI score ranges from 0 to 21, and higher scores indicate worse sleep quality.
ISI (insomnia severity index) | Baseline (week 0) and post-treatment (week 12)
  Changes in ISI scores after 12-week treatment. A total ISI score range from 0 to 28 and categories: 0-7 (No clinically significant insomnia), 8-14 (Subthreshold insomnia), 15-21 (Moderate insomnia), and 22-28 (Severe insomnia)
Johns Hopkins Restless legs syndrome quality of life | Baseline (week 0) and post-treatment (week 12)
  Changes in Johns Hopkins Restless legs syndrome quality of life scores after 12-week treatment. A total score ranges from 0 to 100 and lower scores indicate worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Young Jung, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sunwoo JS, Cho YW, Shin WC, Byun JI, Shin JW, Jung KY. Efficacy and Safety of Pregabalin for Restless Legs Syndrome in Korean Adults: A Randomized, Double-Blind, Placebo-Controlled Trial. J Clin Neurol. 2025 Jul;21(4):325-331. doi: 10.3988/jcn.2025.0092. PMID 40635537